CLINICAL TRIAL: NCT01637493
Title: Safety,Tolerability,Pharmacokinetics and Pharmacodynamics Phase 1 Study of Pegfilgrastim in Chemotherapy Patients
Brief Title: Pharmacokinetics and Pharmacodynamics Study of Pegfilgrastim in Chemotherapy Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Jiuyuan Gene Engineering Co. Ltd., (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY062011A
Record Dates: First submitted 2012-07-02; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Neutropenia
Keywords: Pegylation; G-CSF; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pegfilgrastim, 30mcg/kg (Experimental)
  Interventions: Drug: Pegfilgrastim
- Pegfilgrastim, 60mcg/kg (Experimental)
  Interventions: Drug: Pegfilgrastim
- Pegfilgrastim, 100mcg/kg (Experimental)
  Interventions: Drug: Pegfilgrastim
- Pegfilgrastim, 200mcg/kg (Experimental)
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — Single SC injection of the appropriate dose of drug ranging from 30 mcg/kg to 200 mcg/kg at postchemotherapy 48hr in cycle 2, followed by two doses SC injection of the appropriate dose of drug ranging from 15 mcg/kg to 100 mcg/kg at postchemotherapy 48hr in cycle 3.
  Arms: Pegfilgrastim, 30mcg/kg
Drug: Pegfilgrastim — Single SC injection of the appropriate dose of drug ranging from 30 mcg/kg to 200 mcg/kg at postchemotherapy 48hr in cycle 2, followed by two doses SC injection of the appropriate dose of drug ranging from 15 mcg/kg to 100 mcg/kg at postchemotherapy 48hr in cycle 3.
  Arms: Pegfilgrastim, 60mcg/kg
Drug: Pegfilgrastim — Single SC injection of the appropriate dose of drug ranging from 30 mcg/kg to 200 mcg/kg at postchemotherapy 48hr in cycle 2, followed by two doses SC injection of the appropriate dose of drug ranging from 15 mcg/kg to 100 mcg/kg at postchemotherapy 48hr in cycle 3.
  Arms: Pegfilgrastim, 100mcg/kg
Drug: Pegfilgrastim — Single SC injection of the appropriate dose of drug ranging from 30 mcg/kg to 200 mcg/kg at postchemotherapy 48hr in cycle 2, followed by two doses SC injection of the appropriate dose of drug ranging from 15 mcg/kg to 100 mcg/kg at postchemotherapy 48hr in cycle 3.
  Arms: Pegfilgrastim, 200mcg/kg

SUMMARY:
The purpose of this study is to examine the safety,tolerability,pharmacokinetics and pharmacodynamics of Pegfilgrastim in patients with chemotherapy-induced neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18～70 years
* Confirmed malignant tumor patients by histopathological or cytological diagnosis, not previously treated with chemotherapy or radiotherapy,suitable for chemotherapy with carboplatin combined with taxol or cyclophosphamide combined with pharmorubicin
* Karnofsky score ≥ 70
* Normal coagulation function, no evidences of hemorrhage,WBC ≥ 3,500 per cubic milliliter, ANC ≥ 1,500 per cubic milliliter, PLT ≥ 100,000 per cubic milliliter
* Normal liver, heart, kidney function
* Life expectancy > 3 months
* Signed informed consent

Exclusion Criteria:

* Not adequately controlled infections(e.g. ANC ≥ 12,000 per cubic milliliter,temperature > 38.2℃)
* Evidence of metastatic disease in bone marrow,or with other malignant tumors
* Subjects with symptomatic brain metastases
* Pregnant or breast-feeding or in menstrual period females
* Participated more than 3 clinical trials in nearly a year(as subjects)
* Currently participated in any other clinical trials,or Used any prescription medication could impact on the metabolism of investigational drug, or participated in any other clinical trial within one month from the date of the screening visit
* Donation of whole blood or a unit of blood within three months prior to the start of study
* Known hypersensitivity to filgrastim or any of the products to be administered during dosing
* Evidence of, or treatment for, drug or alcohol abuse within one year from date of screening visit
* Other conditions which in the opinion of the investigator preclude enrollment into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Blood concentration of pegfilgrastim for pharmacokinetics | 42 days

SECONDARY OUTCOMES:
Absolute Neutrophil Count (ANC) | 63 days
CD34+ Cell count | 63 days
Pharmacokinetics: AUC(0-t),Cmax, Tmax, half-life,Cl | 42 days
Safety data: including physical examinations ( include injection site reactions) , laboratory evaluations( ECGs, AST, ALT, Cr, BUN, hemostasis and coagulation test, electrolyte test ), vital signs assessments, and adverse effects (AEs). | 63days
samples for immunogenicity | days 21,42,63

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuankai, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Roskos LK, Lum P, Lockbaum P, Schwab G, Yang BB. Pharmacokinetic/pharmacodynamic modeling of pegfilgrastim in healthy subjects. J Clin Pharmacol. 2006 Jul;46(7):747-57. doi: 10.1177/0091270006288731. PMID 16809800
- [Background] Johnston E, Crawford J, Blackwell S, Bjurstrom T, Lockbaum P, Roskos L, Yang BB, Gardner S, Miller-Messana MA, Shoemaker D, Garst J, Schwab G. Randomized, dose-escalation study of SD/01 compared with daily filgrastim in patients receiving chemotherapy. J Clin Oncol. 2000 Jul;18(13):2522-8. doi: 10.1200/JCO.2000.18.13.2522. PMID 10893282